CLINICAL TRIAL: NCT05497284
Title: A Participant- and Investigator-blinded, Randomized, Placebo-controlled, Multicenter, Platform Study to Investigate Efficacy, Safety, and Tolerability of Various Single Treatments in Participants With Idiopathic Pulmonary Fibrosis
Brief Title: To Assess the Efficacy of the Investigational Products Compared to Placebo in Participants With IPF
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor Decision
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CADPT09A12201
Record Dates: First submitted 2022-08-05; First posted 2022-08-11 (Actual); Results first posted 2025-09-18 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2025-12

CONDITIONS: Idiopathic Pulmonary Fibrosis
Keywords: Idiopathic pulmonary fibrosis; FVC; DLCO; 6-minute walk test; patient reported outcome; HRCT
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- LTP001 (Experimental): LTP001 orally once daily in the morning for approximately 26 weeks.
  Interventions: Drug: LTP001; Drug: Standard of Care (SoC)
- Placebo (Experimental): Placebo orally once daily in the morning for approximately 26 weeks.
  Interventions: Drug: Placebo; Drug: Standard of Care (SoC)

INTERVENTIONS:
Drug: LTP001 — LTP001 administered once daily in the morning
  Arms: LTP001
Drug: Placebo — Placebo to LTP001 administered once daily in the morning
  Arms: Placebo
Drug: Standard of Care (SoC) — nintedanib, pirfenidone, or neither

SUMMARY:
A participant- and investigator-blinded, randomized, placebo-controlled, multicenter, platform study to investigate efficacy, safety, and tolerability of various single treatments in participants with idiopathic pulmonary fibrosis

DETAILED DESCRIPTION:
This was a randomized, placebo-controlled, participant- and investigator-blinded platform study in participants with idiopathic pulmonary fibrosis. Participants underwent a screening period of 42 days, a treatment period of 26 weeks and a post-treatment safety follow-up period of 30 days. This study was designed to safely allow rapid and efficient screening of potentially efficacious investigational products in participants with IPF. The study was terminated for strategic reasons and no additional cohorts were created.

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants at least 40 years of age
* IPF diagnosed based on ATS/ERS/JRS/ALAT IPF 2018 modified guidelines
* FVC ≥45% predicted
* DLCO, corrected for hemoglobin, ≥25% predicted (inclusive)
* Unlikely to undergo lung transplantation during this trial in the opinion of the investigator
* If a participant is taking nintedanib or pirfenidone, they must be on a stable regimen for at least 8 weeks prior to randomization

Exclusion Criteria:

* Airway obstruction (i.e. prebronchodilator FEV1/ FVC < 0.7) or evidence of a bronchodilator response at screening
* Emphysema >20% on screening HRCT
* Fibrosis <10% on screening HRCT
* Clinical diagnosis of any connective tissue disease
* Clinically diagnosed acute exacerbation of IPF (AE-IPF) or other significant clinical worsening within 3 months of randomization

Additional protocol-defined inclusion / exclusion criteria may apply.

Ages: 40 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2022-11-10 (Actual); Primary Completion 2024-08-26 (Actual); Study Completion 2024-09-26 (Actual)

CONTACTS AND LOCATIONS:
Locations (15):
- United States (2):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of Kansas Hospital, Kansas City, Kansas
- Argentina (3):
  - Novartis Investigative Site, CABA, Buenos Aires
  - Novartis Investigative Site, Ranelagh Partido de Berazate, Buenos Aires
  - Novartis Investigative Site, Paraná
- Australia (3):
  - Novartis Investigative Site, Camperdown, New South Wales
  - Novartis Investigative Site, Chermside, Queensland
  - Novartis Investigative Site, Spearwood, Western Australia
- Novartis Investigative Site, Prague, Czechia
- Germany (3):
  - Novartis Investigative Site, Munich, Bavaria
  - Novartis Investigative Site, Coswig
  - Novartis Investigative Site, Essen
- Netherlands (2):
  - Novartis Investigative Site, Amsterdam, North Holland
  - Novartis Investigative Site, Nieuwegein, Utrecht
- Novartis Investigative Site, Bialystok, Poland

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations. This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- See also: A Plain Language Trial Summary is available on www.novctrd.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=2839

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part at 15 investigative sites in 7 countries.
Pre-assignment Details: The screening period took place over 42 days to assess participants eligibility to take part. Written informed consent was obtained from each participant before any study specific proceedure(s) were performed. The study was explained to each participant or designee, who answered and questions, and written information was also provided.
Groups:
- LTP001 6mg: LTP001 6mg orally once daily in the morning for approximately 26 weeks.
Period: Overall Study
Arm/Group | LTP001 6mg | Placebo
Started | 23 | 23
Completed | 15 | 17
Not Completed | 8 | 6
Not completed — Adverse Event | 1 | 0
Not completed — Physician Decision | 0 | 1
Not completed — Study terminated by sponsor | 7 | 4
Not completed — Subject Decision | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | LTP001 6mg | Placebo | Total
Number analyzed (Participants) | 23 | 23 | 46
Age, Continuous [Mean (Standard Deviation); unit: Years] | 70.3 (7.07) | 69.5 (5.34) | 69.9 (6.21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 11 | 13
  Male | 21 | 12 | 33
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 23 | 23 | 46

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to End of Treatment Epoch in Forced Vital Capacity (FVC) Expressed in Percent Predicted
Description: Forced Vital Capacity (FVC) is the total amount of air exhaled during the Forced expiratory volume (FEV) test measured through spirometry testing. FEV measures how much air a person can exhale during a forced breath. It is expressed as percent predicted, defined as FVC of the participant divided by the average FVC in the population for any person of similar age, sex, and body composition multiplied by 100. A positive change from baseline is considered a favorable outcome.
Time Frame: Baseline, up to approximately 26 weeks
Population: The Pharmacodynamic (PD) analysis set included all participants with available PD data and no protocol deviations with relevant impact on PD data. Only participants with evaluable measurements are included.
Measure: Mean (Standard Deviation); unit: Percentage of predicted FVC
Arm/Group | LTP001 6mg | Placebo
Number analyzed (Participants) | 17 | 22
Percentage of predicted FVC | -3.1 (4.80) | -1.1 (5.31)
Statistical Analysis 1: Comparison: LTP001 6mg vs Placebo; Test type: Other — Probability (LTP001 is better than placebo); Baysesian random slope model — Probability that LTP001 is better than placebo is 10.3%; Bayesian random slope model to assess the difference in reduction rate (slope) in years between the treatment group and placebo group; Slope = -2.6, 80% CI 2-sided [-6.9 to 1.3], Standard Deviation 2.07

2. Secondary Outcome: Change From Baseline to End of Treatment Epoch in FVC
Description: Forced Vital Capacity (FVC) is the total amount of air exhaled during the Forced expiratory volume (FEV) test measured through spirometry testing. FEV measures how much air a person can exhale during a forced breath. A positive change from baseline is considered a favorable outcome.
Time Frame: Baseline, up to approximately 26 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | LTP001 6mg | Placebo
Number analyzed (Participants) | 17 | 22
mL | -120.0 (181.56) | -45.5 (176.25)

3. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS is defined as the time from the date of randomization to the date of the any of the following events: Absolute reduction from baseline of ≥10% predicted in FVC, Nonelective hospitalization for respiratory events, Lung Transplant, Death. PFS was analyzed based on Kaplan-Meier estimates.
Time Frame: Baseline, up to approximately 26 weeks
Population: The Pharmacodynamic (PD) analysis set included all participants with available PD data and no protocol deviations with relevant impact on PD data.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | LTP001 6mg | Placebo
Number analyzed (Participants) | 19 | 23
Days | 185.0 [180.0 to NA] — Not estimable due to insufficient number of participants with events. | 185.0 [183.0 to NA] — Not estimable due to insufficient number of participants with events.

4. Secondary Outcome: Number of Participants With Absolute Decline of ≥10% Predicted in FVC
Description: Binary output of absolute decline of ≥ 10% predicted in FVC (Yes/No) at the end of treatment epoch.
Time Frame: Baseline, up to approximately 26 weeks
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | LTP001 6mg | Placebo
Number analyzed (Participants) | 19 | 23
Participants | 6 | 5

5. Secondary Outcome: Change From Baseline to the End of Treatment Epoch in Diffusion Capacity of Lung for Carbon Monoxide (DLCO)
Description: Diffusing capacity of the lungs for carbon monoxide (DLCO) is a measurement to assess the ability of the lungs to transfer gas from inspired air to the bloodstream. Inhaled carbon monoxide (CO) is used for this test due to its high affinity for hemoglobin. During a ten-second breath-hold, DLCO measures uptake of CO per time per CO pressure.
Time Frame: Baseline, up to approximately 26 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mL/min/mmHg
Arm/Group | LTP001 6mg | Placebo
Number analyzed (Participants) | 16 | 17
mL/min/mmHg | -0.167 (1.5568) | -0.334 (2.3838)

6. Secondary Outcome: Change From Baseline to the End of Treatment Epoch in 6-minute Walk Distance (6MWD)
Description: The 6MWD test is self-paced, with standardized instructions and encouragement being given as participants walk as far as possible over 6 minutes through a flat corridor. The final distance is recorded in meters. A positive change from baseline in 6MWD is considered a favourable outcome.
Time Frame: Baseline, up to approximately 26 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | LTP001 6mg | Placebo
Number analyzed (Participants) | 14 | 20
meters | 9.2 (63.06) | 4.7 (56.66)

7. Secondary Outcome: Change From Baseline to the End of Treatment Epoch in Total Score From the K-BILD Questionnaire
Description: The King's Brief Interstitial Lung Disease (K-BILD) is a 15-item HRQOL questionnaire that range from 0 to 100. Higher scores indicate better health-related quality of life, with 100 representing the best possible health status. A positive change from baseline in K-BILD questionnaire is considered a favourable outcome.
Time Frame: Baseline, up to approximately 26 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | LTP001 6mg | Placebo
Number analyzed (Participants) | 17 | 22
score on scale | 17.17 (174.009) | 7.94 (136.768)

8. Secondary Outcome: Change From Baseline to the End of Treatment Epoch in Scores From Leicester Cough Questionnaire
Description: The Leicester Cough Questionnaire (LCQ) is a 19-item validated patient-report questionnaire that measures the impact of cough on quality of life. It takes about 5 minutes to complete and results in three domain scores (Social, Psychological, and Physical), and one Total score. Domain scores are averages of the questions that make up each domain. Minimum and maximum domain scores are 1 and 7, respectively. The domain scores are summed to determine the Total score, which can range from 3 to 21. A higher score means less impact on quality of life. A positive LCQ change score indicates an improvement.
Time Frame: Baseline, up to approximately 26 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | LTP001 6mg | Placebo
Number analyzed (Participants) | 17 | 22
score on scale | -3.9 (14.23) | 2.7 (18.35)

9. Secondary Outcome: Change From Baseline to the End of Treatment Epoch in Scores From the the R-Scale for IPF Questionnaire
Description: The Raghu-Scale for Pulmonary Fibrosis (R-Scale for PF) is a questionnaire designed to assess the impact of lung disease on quality of life. The R-Scale-PF uses a numerical rating scale to assess the severity of five symptoms: cough, shortness of breath, fatigue, depressed mood, and overall sense of wellbeing, over the past two weeks. Each item is scored from 0 to 10, with lower scores indicating better health-related quality of life. The total R-Scale-PF score ranges from 0 to 50. A decrease from baseline in R-Scale for PF is considered a favourable outcome.
Time Frame: Baseline, up to approximately 26 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | LTP001 6mg | Placebo
Number analyzed (Participants) | 17 | 22
score on scale | 1.53 (5.784) | -0.93 (6.020)

10. Secondary Outcome: Change From Baseline to the End of Treatment Epoch in Total Score From the Living With IPF Questionnaire
Description: Living with idiopathic pulmonary fibrosis (L-IPF) is a tool that assesses symptoms and impacts of IPF. The Symptoms Module consists of 20 questions to assess symptoms experienced from IPF over the last 24 hours. The Impacts Module consists of 20 questions on how IPF affects quality of life over the last 7 days. The total score ranging from 0 to 100, with higher scores indicating greater symptom severity. A positive change from baseline in L-IPF is considered a favourable outcome.
Time Frame: Baseline, up to approximately 26 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | LTP001 6mg | Placebo
Number analyzed (Participants) | 17 | 22
score on scale | 7.15 (14.392) | -4.48 (11.067)

ADVERSE EVENTS:
Time Frame: Adverse events were reported from first dose of study treatment until end of study treatment plus follow up period, up to a maximum duration of approximately 30 weeks.
Groups:
- LTP001 6 mg: LTP001 6mg orally once daily in the morning for approximately 26 weeks.
- Total: Total
Arm/Group | LTP001 6 mg | Placebo | Total
All-Cause Mortality (participants affected / at risk) | 1/23 | 0/23 | 1/46
Serious Adverse Events (participants affected / at risk) | 2/23 | 1/23 | 3/46
Other Adverse Events (participants affected / at risk) | 14/23 | 7/23 | 21/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LTP001 6 mg (N=23) | Placebo (N=23) | Total (N=46)
Herpes zoster (Infections and infestations) | 1 | 0 | 1
Infection (Infections and infestations) | 1 | 0 | 1
Bladder disorder (Renal and urinary disorders) | 1 | 0 | 1
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | LTP001 6 mg (N=23) | Placebo (N=23) | Total (N=46)
Diarrhoea (Gastrointestinal disorders) | 5 | 1 | 6
Bronchitis (Infections and infestations) | 2 | 0 | 2
Pneumonia (Infections and infestations) | 0 | 2 | 2
Urinary tract infection (Infections and infestations) | 1 | 2 | 3
Amylase increased (Investigations) | 2 | 0 | 2
Lipase increased (Investigations) | 2 | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 1 | 4
Headache (Nervous system disorders) | 1 | 2 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 3
Hypertension (Vascular disorders) | 2 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2023-10-09): https://cdn.clinicaltrials.gov/large-docs/84/NCT05497284/Prot_000.pdf
  • Statistical Analysis Plan (2024-11-12): https://cdn.clinicaltrials.gov/large-docs/84/NCT05497284/SAP_001.pdf